CLINICAL TRIAL: NCT00505154
Title: A Phase III Study of the Effect of Rosuvastatin on Left Ventricular Remodeling and Inflammatory Markers in Heart Failure
Brief Title: Effect of Rosuvastatin on Left Ventricular Remodeling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Gullestad, Professor, Rikshospitalet University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG012007
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Dilated Cardiomyopathy
Keywords: Heart failure; inflammation; cytokines
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Inflammation | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo tablets
  Interventions: Drug: placebo
- 1 (Active Comparator): rosuvastatin
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 10 mg tablets od for 6 months
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to examine the the effect of the HMG-CoA reductase inhibitor Rosuvastatin on left ventricular remodeling in patients with dilated cardiomyopathy.

DETAILED DESCRIPTION:
* Chronic heart failure (HF) is one of the most important public health problems in cardiovascular medicine.
* Idioatic dilated cardiomyopathy (CMP) represents the final common expression of primary myocardial damage produced by a variety of as yet undefined myocardial insults, producing areas of interstitial and perivascular fibrosis, particularly of the left ventricle. Chronic HF, including CMP, is a progressive disease with high morbidity and mortality, suggesting that important pathogenic mechanisms remain active and unmodified by the present treatment modalities. The presence of chronic inflammation in patients with chronic heart failure has been widely recognized and coupled with persistent immune activation may represent such unmodified mechanisms.

The effect of statin therapy on lipids are well known, but recent studies suggest that the beneficial effects of statins also may be related to their anti-inflammatory properties.

To further elucidate this issue we want to study the potent new statin Rosuvastatin on myocardial function and remodeling and their relation to inflammatory markers in patients with IDCM. As hyperlipidemia is not involved in the pathogenesis of IDCM, as opposed to HF secondary to CAD, such studies will also be an interesting approach in separating the lipid lowering from other effects of these medications in HF.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-80 years
* Have clinical or symptomatic evidence of HF, in NYHA class II-IV, for at least 3 months
* Have LVEF <40%
* On optimal medical treatment and considered unsuitable for surgical intervention.
* Have given written informed consent
* No planned heart transplantation
* Female of potential childbearing age must have a negative serum pregnancy test within 7 days prior to enrollment. Effective contraception must be used during the trial and for 6 weeks following discontinuation of the study medication, even where there has been a history of infertility.

Exclusion Criteria:

* Evidence of unstable disease
* Evidence of ischemic etiology on the basis of history (diagnosed myocardial infarction), echocardiography or angiography)
* Evidence of clinical significant valvular disease based on echocardiography
* Significant concomitant diseases such as infections, pulmonary disease or connective tissue disease.
* Contraindication against statin therapy

  * Hypersensitivity against statins
  * Liver disease with SGOT and SGPT > 2 timer upper normal limit
  * Baseline elevations of CK 3 times upper normal values at any time during the course of the study
  * Serum creatinine above 2.0 mg/dL (177 umol/L) at any time during the course of the study
  * Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
End points will be LV end systolic and diastolic volume (LVESV, LVEDV), and LV-ejection fraction (LV-EF). | 2009

SECONDARY OUTCOMES:
the B-type natriuretic peptide (BNP), Effect on immunological variables | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Geir Gokstad, Study Director — Rikshospitalet, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Broch K, Askevold ET, Gjertsen E, Ueland T, Yndestad A, Godang K, Stueflotten W, Andreassen J, Svendsmark R, Smith HJ, Aakhus S, Aukrust P, Gullestad L. The effect of rosuvastatin on inflammation, matrix turnover and left ventricular remodeling in dilated cardiomyopathy: a randomized, controlled trial. PLoS One. 2014 Feb 25;9(2):e89732. doi: 10.1371/journal.pone.0089732. eCollection 2014. PMID 24586994